CLINICAL TRIAL: NCT01790815
Title: Mothers Understand And Can do it - Mid Upper Arm Circumference Screening for Malnutrition Performed by Mothers of Children < 5 Years Old
Brief Title: Mothers Understand And Can do it - Mid Upper Arm Circumference Screening for Malnutrition Performed by Mothers
Acronym: MUAC
Status: Completed | Type: Observational
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Bien Être de La femme et de L'Enfant au Niger (Unknown)
Responsible Party: Sponsor
Other Study IDs: MUAC mères
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Marasmus; Kwashiorkor; Malnutrition; Degree, Moderate; Malnutrition
Keywords: Acute Malnutrition; Mid Upper Arm Circumference; Screening
MeSH Terms: conditions — Protein-Energy Malnutrition; Kwashiorkor; Malnutrition; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
PRIMARY OBJECTIVE :

To determine whether mothers, given minimal group training, are capable of using a MUAC (mid-upper arm circumference) bracelet to screen their children for malnutrition and categorise them into one of three groups : 'red' (SAM ; severe acute malnutrition), 'yellow' (MAM ; moderate acute malnutrition) or 'green' (normal nutritional status)

SECONDARY OBJECTIVES :

To establish whether there is a difference in the MUAC value if measured on the right arm as opposed to the left, in young children

To determine whether there is a difference in the MUAC value if the mid upper arm position is determined visually as opposed to being measured in the 'classical' fashion

DETAILED DESCRIPTION:
Severe Acute Malnutrition (SAM) and its complications are major causes of death in under 5s in the developing world. A simple, reproducible, scalable way to recognise acute malnutrition and target early intervention would be a huge advance. Can mothers with limited training reliably measure and interpret the results of Mid Upper Arm Circumference (MUAC), a measurement performed with a MUAC measuring tape costing $0.06? MUAC contrasts with Z-score (WHZ), which requires both scales and a height gauge, both health worker interventions susceptible to considerable error, sensitive to non-nutritional factors, requiring calculations and growth curves, yet much less accurate in predicting risk of death compared with MUAC.

ELIGIBILITY:
Inclusion Criteria:

* children present in the inpatient malnutrition treatment unit and paediatric service of the Mirriah district hospital aged between 6-59 months old
* children aged between 6-59 months old in the two villages where the community phase of the study was conducted

Exclusion Criteria:

* children receiving treatment in the intensive care unit of Mirriah district hospital
* children with bilateral oedema
* children whose mothers or fathers refused consent to participate in the study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children present in the inpatient malnutrition treatment unit and paediatric service of the Mirriah district hospital aged between 6-59 months old
  Children aged between 6-59 months old in the two villages of the Mirriah district, Niger; where the community phase of the study was conducted
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
inter and intra observer variability | 2 years
  Variance in result of screening for malnutrition performed by mothers with minimal training compared to 'gold-standard' fully trained health care workers. Screening will be performed with a MUAC (mid-upper arm circumference) bracelet, results will be expressed by category: SAM (severe acute malnutrition), MAM (moderate acute malnutrition) or 'normal nutritional status

SECONDARY OUTCOMES:
inter and intra observer variability | 2 years
  The difference in millimetres in the MUAC value if measured on the right arm as opposed to the left ('classical method'), in young children
inter and intra observer variability | 2 years
  The difference in the MUAC value in millimetres if the mid upper arm position is determined visually as opposed to being measured in the 'classical' fashion

CONTACTS AND LOCATIONS:
Overall Officials: nikki blackwell, FCICM,FRACP, Study Director — Alliance for International Medical Action
Locations (1):
- Mirriah Health District, Mirriah, Mirriah, Niger

REFERENCES:
- [Background] Briend A, Maire B, Fontaine O, Garenne M. Mid-upper arm circumference and weight-for-height to identify high-risk malnourished under-five children. Matern Child Nutr. 2012 Jan;8(1):130-3. doi: 10.1111/j.1740-8709.2011.00340.x. Epub 2011 Sep 28. PMID 21951349
- [Background] Briend A, Garenne M, Maire B, Fontaine O, Dieng K. Nutritional status, age and survival: the muscle mass hypothesis. Eur J Clin Nutr. 1989 Oct;43(10):715-26. PMID 2612460
- [Derived] Blackwell N, Myatt M, Allafort-Duverger T, Balogoun A, Ibrahim A, Briend A. Mothers Understand And Can do it (MUAC): a comparison of mothers and community health workers determining mid-upper arm circumference in 103 children aged from 6 months to 5 years. Arch Public Health. 2015 May 18;73(1):26. doi: 10.1186/s13690-015-0074-z. eCollection 2015. PMID 25992287
- See also: Click here for more information about the Alliance for International Medical Action — http://www.alimaong.org